CLINICAL TRIAL: NCT02923739
Title: A Randomized Phase II Induction Discontinuation Trial of Emactuzumab Following Paclitaxel and Bevacizumab in Patients With Platinum-Resistant, Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Paclitaxel and Bevacizumab With or Without Emactuzumab in Treating Patients With Platinum-Resistant Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by the Sponsor
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0647; NCI-2016-01593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0647 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-09-30; First posted 2016-10-05 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fallopian Tube Adenocarcinoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Mucinous Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Fallopian Tube Transitional Cell Carcinoma; Fallopian Tube Undifferentiated Carcinoma; Malignant Ovarian Brenner Tumor; Ovarian Adenocarcinoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Mucinous Adenocarcinoma; Ovarian Seromucinous Carcinoma; Ovarian Serous Adenocarcinoma; Ovarian Transitional Cell Carcinoma; Ovarian Undifferentiated Carcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Brenner Tumor; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; emactuzumab; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (paclitaxel, bevacizumab) (Active Comparator): Patients receive paclitaxel IV over 60 minutes on days 1, 8, 15, and 22 and bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel
- Arm II (paclitaxel, bevacizumab, emactuzumab) (Experimental): Patients receive paclitaxel and bevacizumab as in Arm I. Patients also receive emactuzumab IV over 30 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Biological: Emactuzumab; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Pharmacological Study

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; BEVACIZUMAB, LICENSE HOLDER UNSPECIFIED; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Biological: Emactuzumab — Given IV
  Other Names: RG-7155; RG7155; RO-5509554; RO5509554
  Arms: Arm II (paclitaxel, bevacizumab, emactuzumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Pharmacological Study — Correlative studies
  Arms: Arm II (paclitaxel, bevacizumab, emactuzumab)

SUMMARY:
This randomized phase II trial studies the side effects of paclitaxel and bevacizumab with or without emactuzumab and how well they work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back after treatment with platinum chemotherapy. Monoclonal antibodies, such as emactuzumab, block tumor growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Bevacizumab may prevent the growth of new blood vessels that tumors need to grow. Giving emactuzumab with paclitaxel and bevacizumab may work better in treating ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety of administration of paclitaxel, bevacizumab and emactuzumab over 4 weeks. (Part 1) II. To compare the progression-free survival (PFS) of patients with stable disease following Part 2A randomized to paclitaxel plus bevacizumab or to paclitaxel, bevacizumab plus emactuzumab. (Part 2B)

SECONDARY OBJECTIVES:

I. To estimate the progression-free survival (PFS) of the treatment arms. II. Objective response rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) and CA-125 response criteria ("responders").

III. Objective response rate by RECIST only ("RECIST responders"). IV. Objective response rate by CA-125 response criteria only ("CA-125 responders").

V. Biological progression-free interval (PFIbio) by serum CA-125 assessed according to the Gynecologic Cancer Intergroup (GCIG) criteria.

VI. Overall survival (OS). VII. Safety and tolerability. VIII. To characterize the pharmacokinetics of bevacizumab and emactuzumab when administered in combination.

EXPLORATORY OBJECTIVES:

I. To assess the utility of surrogate biomarkers and the anti-tumor response to therapy with the combination treatment of bevacizumab and emactuzumab.

II. To assess tumor alterations by serial non-invasive imaging macrophage-specific imaging, ADC (apparent diffusion coefficient) for cellularity, and DCE (dynamic contrast enhanced) for vasculature.

OUTLINE:

Patients receive paclitaxel intravenously (IV) over 60 minutes on days 1, 8, 15, and 22 and bevacizumab IV over 90 minutes on days 1 and 15. Treatment repeats every 28 days for up to 2 courses in the absence of disease progression or unexpected toxicity. Patients with stable disease are randomized to 1 of 2 arms.

ARM I: Patients receive paclitaxel IV over 60 minutes on days 1, 8, 15, and 22 and bevacizumab IV over 90 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive paclitaxel and bevacizumab as in Arm I. Patients also receive emactuzumab IV over 30 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, every 3 months for 2 years, every 4 months for 1 year, and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the study requirements (inclusive of 2 biopsies, one at baseline and if they qualify, one pre-randomization for part 2B)
* Women 18 years of age or older
* Histologically confirmed and documented disease to include: adenocarcinoma NOS (not otherwise specified), clear cell adenocarcinoma, endometrioid adenocarcinoma, malignant Brenner's tumor, mixed epithelial carcinoma, mucinous adenocarcinoma, serous adenocarcinoma, transitional cell carcinoma, and undifferentiated carcinoma
* Patients must have platinum-resistant disease, (defined as progression within < 6 months from completion of a minimum of 4 platinum therapy cycles (+ 7 days); the date should be calculated from the last administered dose of platinum therapy)
* Patients must have disease that is measurable according to RECIST 1.1 or assessable according to the GCIG CA-125 criteria and require chemotherapy treatment; part 1: patients must have one or more measurable target lesion; part 2: patients must have two or more measurable target lesions; measurable disease is defined at least one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded); each 'target' lesion must be >= 20 mm when measured by conventional techniques, including palpation, plain x-ray, computed tomography (CT), and magnetic resonance imaging (MRI), or >= 10 mm when measured by spiral CT
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Newly obtained core or excisional biopsy of a tumor lesion for part 2A and if they qualify, one pre-randomization biopsy for part 2B
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Hemoglobin >=9 g/dL or >= 5.6 mmol/L
* Creatinine clearance >= 60 mL/min for subject with creatinine levels > 1.5 X institutional upper limit of normal (ULN)
* Total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGOT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* International normalized ratio (INR)/prothrombin time (PT) =< 1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time [PTT] is within therapeutic range of intended use of anticoagulants)
* PTT =< 1.5 X ULN (unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
* Life expectancy of >= 12 weeks

Exclusion Criteria:

* Patients who have disease progression prior to completion of intended frontline therapy, including patients demonstrating disease progression after interval cytoreduction
* Non-epithelial, including malignant mixed Mullerian tumors
* Ovarian tumors with low malignant potential (i.e. borderline tumors)
* For part 2 patients only: History of other clinically active malignancy within 5 years of enrollment, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal-cell carcinoma or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix or breast, or early stage endometrial cancer (stage IA/B, grade 1 or 2, endometrioid histology)
* Previous treatment with > 2 anticancer regimens for ovarian cancer
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment, with the following exceptions: hormone-replacement therapy or oral contraceptives; tyrosine kinase inhibitors (TKIs) that have been discontinued > 7 days prior to cycle 1, day 1; screening scans must be obtained after discontinuation of prior TKIs
* Any prior radiotherapy to the pelvis or abdomen
* Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to study enrollment, or anticipation of need for major surgical procedure during the course of the study; minor surgical procedures including placement of a vascular access device, within 2 days of the first study treatment
* Previous exposure to murine CA-125 antibody (only applicable to those patients with non-measurable disease by RECIST)
* Current or recent (within 10 days prior to the first study drug dose) chronic daily treatment with aspirin (> 325 mg/day)
* Current or recent treatment with another investigational drug within 30 days of first study treatment dosing or earlier participation in this study
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents within 2 weeks prior to cycle 1, day 1; patients who have received acute and/or lowrolment, or anticipation of need for major surgical, a one-time dose of dexamethasone for nausea or chronic use of =< 10 mg/day of prednisone or dose-equivalent corticosteroid) may be enrolled in the study after discussion with and approval by the medical monitor; the use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed; prior corticosteroids as anti-cancer therapy within a minimum of 14 days of first receipt of study drug
* Received therapeutic oral or IV antibiotics within 2 weeks prior to cycle 1, day 1; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Patients with urine dipstick for proteinuria > 2+; patients with >= 2+ proteinuria on baseline dipstick analysis should undergo a 24-hour urine collection and must demonstrate =< 1 g of protein in the 24-hour urine; alternatively, proteinuria testing can be performed according to local standards
* Patients with known auto-immune disease
* Patients with known history of human immunodeficiency virus (HIV), hepatitis B virus (HBV) and hepatitis C virus (HCV) infection
* Patient has received an organ transplant
* Patient has a history of hematological malignancy within the last 5 years prior to study entry; prior allogeneic bone marrow transplantation or prior solid organ transplantation
* Patient has a history of hematological malignancy within the last 5 years prior to study entry
* History of or active autoimmune disease including, but not limited to, systemic lupus erythematous, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, and vasculitis or glomerulonephritis; patients with autoimmune thyroid disease on a stable thyroid replacement regimen; controlled vitiligo, eczema, psoriasis, or seborrheic dermatitis with only dermatologic manifestations; or controlled type I diabetes on a stable insulin regimen may be eligible for the study with approval by the medical monitor
* History or evidence upon physical/neurological examination of central nervous system (CNS) disease unrelated to cancer, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures)
* Symptomatic CNS metastasis
* Pre-existing peripheral neuropathy >= Common Terminology Criteria (CTC) grade 2 for those patients who received prior paclitaxel
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >= 2 weeks prior to screening
* Increased corrected QT (QTc) interval (QTc > 470 ms), patients with baseline resting bradycardia < 45 beats per minute (bpm), or baseline resting tachycardia > 100 bpm
* Family history of long QT syndrome or other risk factors for torsades de pointes, and/or the use of concomitant medications that prolong the QT/QTc interval
* Signs or symptoms of serious active infection requiring oral or i.v. antibiotics within 2 weeks prior to cycle 1 day 1 and/or hospitalization at study entry including, but not limited to, hospitalization for complications of infection, bacteremia, active tuberculosis or severe pneumonia
* Pregnant or lactating females; serum pregnancy test to be assessed within 7 days prior to study treatment start, or within 14 days (with a confirmatory urine pregnancy test within 7 days prior to study treatment start)
* For women who are not postmenopausal (< 12 months of non therapy-induced amenorrhea, with no identified cause other than menopause) and have not undergone surgical sterilization (removal of ovaries and/or uterus): agreement to remain abstinent (refrain from heterosexual intercourse) or use two adequate non hormonal methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 4 months after the last dose of study drug
* Examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, established, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices; the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* History or evidence of thrombotic or hemorrhagic disorders; including cerebrovascular accident (CVA)/stroke or transient ischemic attack (TIA) or sub-arachnoid hemorrhage within =< 6 months prior to the first study treatment
* Uncontrolled hypertension (sustained systolic > 150 mmHg and/or diastolic > 100 mmHg despite antihypertensive therapy) or clinically significant (i.e. active) cardiovascular disease, including: myocardial infarction or unstable angina within =< 6 months prior to the first study treatment; New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF); serious cardiac arrhythmia requiring medication (with the exception of atrial fibrillation or paroxysmal supraventricular tachycardia); significant vascular disease (e.g., aortic aneurysm, requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior of study enrollment; prior history of hypertensive crisis or hypertensive encephalopathy
* History of bowel obstruction, including sub-occlusive disease, related to the underlying disease and history of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess; evidence of recto-sigmoid involvement by pelvic examination or bowel involvement on CT scan or clinical symptoms of bowel obstruction
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* History of hemoptysis (>= 1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment for any tumor type
* Non-healing wound, ulcer or bone fracture
* Known hypersensitivity to any of the study drugs or excipients
* Evidence of any other medical conditions (such as psychiatric illness, peptic ulcer, etc.), physical examination or laboratory findings that may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-05-05 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anil K. Sood, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (8):
- United States (8):
  - MD Anderson Cancer Center at Cooper-Voorhees, Voorhees Township, New Jersey
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - The Woman's Hospital of Texas, Houston, Texas
  - MD Anderson Regional Care Center-Katy, Houston, Texas
  - MD Anderson Regional Care Center-Bay Area, Nassau Bay, Texas
  - MD Anderson Regional Care Center-Sugar Land, Sugar Land, Texas
  - MD Anderson Regional Care Center-The Woodlands, The Woodlands, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 05/05/2017 and closed to new patient entry on 11/19/2018. The study was terminated on 09/27/2022 and all recruitment was done in a medical clinic setting.
Groups:
- Safety Lead-In; Randomized Arm 2: Paclitaxel 80 mg/m2 IV given on Days 1, 8, 15, & 22 plus Bevacizumab 10 mg/Kg IV on Days 1 & 15, and Emactuzumab 1000 mg IV on Days 1 & 15 on a 28 day cycle
- Induction Arm; Randomized Arm 1: Paclitaxel 80 mg/m2 IV given on Days 1, 8, 15, & 22 plus Bevacizumab 10 mg/Kg IV on Days 1 & 15 on a 28 day cycle
Period: Overall Study
Arm/Group | Safety Lead-In | Induction Arm | Randomized Arm 1 | Randomized Arm 2
Started | 9 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Failed Screening | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated early by the sponsor
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Lead-In | Induction Arm | Randomized Arm 1 | Randomized Arm 2 | Total
Number analyzed (Participants) | 9 | 0 | 0 | 0 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 0 | 0 | 5
  >=65 years | 4 | 0 | 0 | 0 | 4
Age, Continuous [Mean (Full Range); unit: Years] | 66 [51 to 77] |  |  |  | 66 [51 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 0 | 0 | 0 | 9
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 0 | 3
  Not Hispanic or Latino | 6 | 0 | 0 | 0 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 7 | 0 | 0 | 0 | 7
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 9 |  |  |  | 9

OUTCOME MEASURES:

1. Primary Outcome: Part 1: To Evaluate the Safety of Administration of Paclitaxel, Bevacizumab and Emactuzumab Over 4 Weeks.
Description: Safety is defined as no required dose alterations during the first cycle (4 weeks) of therapy due to a grade 3 or greater related adverse event.
Time Frame: Up to 4 weeks
Population: The study was terminated early by the sponsor and no data was collected for the study objective was unable to be fully evaluated.
Arm/Group | Safety Lead-In | Induction Arm | Randomized Arm 1 | Randomized Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Primary Outcome: Part 2B: To Compare the Progression-free Survival (PFS) of Patients With Stable Disease Following Part 2A Randomized to Paclitaxel Plus Bevacizumab or to Paclitaxel, Bevacizumab Plus Emactuzumab.
Description: Will use a log-rank test.
Time Frame: At 32 weeks
Population: The study was terminated early by the sponsor and the study objective was unable to be fully evaluated
Arm/Group | Safety Lead-In | Induction Arm | Randomized Arm 1 | Randomized Arm 2
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: The study was terminated early by the sponsor and the study objective was unable to be fully evaluated
Arm/Group | Safety Lead-In | Induction Arm | Randomized Arm 1 | Randomized Arm 2
All-Cause Mortality (participants affected / at risk) | 5/9 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 4/9 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 4/9 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-In (N=9) | Induction Arm (N=0) | Randomized Arm 1 (N=0) | Randomized Arm 2 (N=0)
CPK increased (Investigations) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Lead-In (N=9) | Induction Arm (N=0) | Randomized Arm 1 (N=0) | Randomized Arm 2 (N=0)
LDH increased (Investigations) | 4 (14) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopcia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (16) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SGOT increased (Investigations) | 4 (13) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CPK increased (Investigations) | 4 (18) | 0 (0) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear and labyrinth disorders (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema - face (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - conjunctival chemosis (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (21) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palmar-plantar erythodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT02923739/Prot_SAP_000.pdf